CLINICAL TRIAL: NCT05397977
Title: Comparison of the Effects of Mechanical Traction and Manual Traction on Pain, Muscle Tone and Functionality in Persons With Cervicogenic Headache
Brief Title: Comparison of the Effects of Mechanical Traction and Manual Traction on Cervicogenic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/2021.K-85
Record Dates: First submitted 2022-04-26; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Cervicogenic Headache
Keywords: Traction, Muscle Tone, Headache, Cervicogenic Pain
MeSH Terms: conditions — Post-Traumatic Headache; Headache | interventions — Transcutaneous Electric Nerve Stimulation; Ultrasonography; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mechanical traction group (Experimental): use of device chattanooga tru trac
  Interventions: Device: mechanical traction group
- manual traction group (Active Comparator): use of manual traction with physiotherapist hands
  Interventions: Other: manuel traction group

INTERVENTIONS:
Device: mechanical traction group — In the mechanical traction group, 26 people with cervicogenic headache will be traction with the Chattanooga Tru Trac traction device, 6 days a week for 2 weeks.
  Persons to be mechanically traction will be placed on their backs on the treatment bed with their necks on the neck collar of the device. After the patients are fixed to the head, the pulling force of the device will start with 10% of the patient's body weight, the device will be set as 60 seconds of pulling force and 20 seconds of relaxation. In subsequent sessions, the pulling force will be gradually adjusted based on the patient's previous traction therapy, tolerance, and symptom response. Each session will take 15 minutes.
  Participants will be given 20 minutes of TENS, 20 minutes of hotpack and 4 minutes of ultrasound, and the exercise will be given as a home program.
  Other Names: TENS; ultrasound; hotpack; home exercise programme
  Arms: mechanical traction group
Other: manuel traction group — Manual traction, one of Cyriax's neck mobilization techniques, will be applied to the MTG. Vertebrobasilar artery test will be applied to the patients before starting the treatment, and manual traction will be applied to the patients in case the vertebrobasilar artery test is negative. Manual traction technique will be applied to the cervical region for 15 minutes. While applying manual traction, the patient will be placed on his back with his head hanging off the bed. Grasp the occiput with one hand and under the chin with the other. Manual traction will be applied by keeping the neck neutral and the occiput slightly extended. After applying traction for a few seconds, it will be slowly released and returned to the starting position, and the application will be made for 15 minutes.
  20 minutes of TENS, 20 minutes of hotpack and 4 minutes of ultrasound will be applied to the participants, and the exercise will be given as a home program.
  Other Names: TENS; ultrasound; hotpack; home exercise programme
  Arms: manual traction group

SUMMARY:
52 people between the ages of 18-45 who were diagnosed with cervicogenic headache by the physician who applied to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital will be included in the research. 52 people will be randomized. They will be divided into two groups, 26 people in the study group and 26 people in the control group. The study group will be called the mechanical traction group (CTG), and the control group will be called the manual traction group (MTG).

After obtaining the demographic information of the individuals to be included in the study, the cases will be evaluated with the visual analogue scale (VAS) and Mc-Gill Melzack Pain Questionnaire for head and neck pain before and after treatment. Cervical joint range of motion will be measured with an electrogoniometer, and muscle tone will be measured with myotonometer (MyotonPRO). Flexion and extension endurance tests will be performed on the cervical region muscles. Headache Impact Scale (HIT-6) will be performed to evaluate the functional status of the patients. Posture of patients will be evaluated with Corbin Posture Analysis. Pittsburgh Sleep Quality Index will be used to evaluate the sleep quality of the patients. All patients will be informed about the study. An informed consent form will be obtained from each.

The mechanical traction group (CTG) and the manual traction group (MTG) will be treated for 6 days and 2 weeks.

Intermittent traction with chattanooga tru trac traction device will be applied to CTG, and manual traction, one of Cyriax's neck mobilization techniques, will be applied to MTG.transcutaneous electrical nerve stimulation (TENS), hotpack and ultrasound will be applied to both groups, and an exercise program will be given in the form of a home program.

DETAILED DESCRIPTION:
Cervicogenic headache (CGH) is a unilateral chronic pain that begins in the neck and neck and radiates to the back of the head. Pain in the CGH originates from structures in the cervical region innervated by the C1-C3 spinal nerves. Therefore, possible causes of CGH: Art. atlantooccipital, art. atlantoaxialis, C2-C3 art. It is related to dysfunctions arising from zygapophysial , C2-C3 discus intervertebral, upper cervical spinal nerves and their roots, skeletal muscles, connective tissue and neurovascular structures in the region.

The aim of this study was to compare the effects of mechanical traction and manual traction on pain, muscle tone and functionality in cervicogenic headache.

52 people between the ages of 18-45 who were diagnosed with cervicogenic headache by the physician who applied to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital will be included in the research. 52 people will be randomized. They will be divided into two groups, 26 people in the study group and 26 people in the control group. The study group will be called the mechanical traction group (CTG), and the control group will be called the manual traction group (MTG).

After obtaining the sociodemographic information of the individuals to be included in the study, the patients will be evaluated with the visual analogue scale (VAS) and Mc-Gill Melzack Pain Questionnaire for head and neck pain before and after treatment. Cervical joint range of motion will be measured with an electrogoniometer, and muscle tone will be measured with myotonometer (MyotonPRO). Flexion and extension endurance tests will be performed on the cervical region muscles. Headache Impact Scale (HIT-6) will be performed to evaluate the functional status of the patients. Posture of patients will be evaluated with Corbin Posture Analysis. Pittsburgh Sleep Quality Index will be used to evaluate the sleep quality of the patients. All patients will be informed about the study. An informed consent form will be obtained from each.

The mechanical traction group (CTG) and the manual traction group (MTG) will be treated for 6 days and 2 weeks.

Intermittent traction will be applied to CTG with the chattanooga tru trac traction device. They will be placed on the treatment bed on their back with their necks on the neck collar of the device. After the patients are fixed from the head, the device will be adjusted so that the pulling force of the device starts with 10% of the patients' body weight. The device will be set as 60 seconds of pulling force and 20 seconds of relaxation. Patients will be told that they should feel moderately strong or strong so that the pulling force does not increase symptoms. In the following sessions, the pulling force will be adjusted gradually according to the patient's previous traction treatment, tolerance and symptom response. Each session will last 15 minutes.

Manual traction, one of Cyriax's neck mobilization techniques, will be applied to the MTG. Vertebrobasilar artery test will be applied to the patients before starting the treatment, and manual traction will be applied to the patients in case the vertebrobasilar artery test is negative. Manual traction technique will be applied to the cervical region for 15 minutes. While applying manual traction, the patient will be placed on his back with his head hanging off the bed. Grasp the occiput with one hand and under the chin with the other. Manual traction will be applied by keeping the neck neutral and the occiput slightly extended. After applying traction for a few seconds, it will be slowly released and returned to the starting position, and the application will be made for 15 minutes.

Both groups will be given conventional treatment. In conventional treatment, TENS, hotpack and ultrasound will be performed on patients. TENS treatment will be applied using 4 adhesive electrodes measuring 5 x 5 cm. Cervical paravertebral region, 80 Hz frequency and 180 ms current were used and will be applied for 20 minutes. The current intensity that the patient can feel intensely will be adjusted. Hotpack hot application will be applied for 20-30 minutes. Ultrasound will be applied bilaterally to the cervical paravertebral region with the help of ultrasound gel at 1 megahertz (MHz) and 1.5 W/cm² for 4 minutes, with the ultrasound head in contact with the skin.

Craniocervical flexion exercises, chin tuck, scapular depression and retraction exercises will be given to both groups as a home program.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-45
* having neck or headache for at least 3 months meets the diagnostic criteria for cervicogenic headache.

  1. Unilateral pain
  2. Decreased neck range of motion
  3. Ipsilateral shoulder discomfort
  4. Ipsilateral arm discomfort
  5. Pain increase with different neck movements and pain with palpation eligible persons will be included.

Exclusion Criteria:

* migraine
* cluster headache
* cervical radiculopathy,
* entrapment neuropathy,
* myelopathy,
* rheumatoid arthritis,
* undergo cervical spinal surgery,
* to be pregnant,
* have a whiplash injury
* those who received physical therapy within 6 months will not be included in the study.
* In cases where mechanical traction is contraindicated (inflammatory joint diseases, osteoporosis, acute inflammatory conditions, acute strain and injury, vertebrobasilar artery failure of the circulation, such as stroke or transient ischemic attack. abnormal upper motor neuron lesions, cardiovascular diseases, malignant tumoral conditions) will not be included.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-26 (Estimated)

PRIMARY OUTCOMES:
sociodemographic information change | At baseline
  The sociodemographic information, education level, existence of problems of the individuals participating in the study will be questioned and recorded.
visual analogue scale (VAS) change | change from baseline the visual analogue scale at 2 weeks
  In the evaluation made with VAS, patients will be asked to mark their pain intensity on a 10 cm horizontal line. Ranges for pain intensity; <3 mild pain, 3-6 moderate pain, >6 severe pain
Mc-Gill Melzack Pain Questionnaire change | change from baseline Mc-Gill Melzack Pain Questionnaire at 2 weeks
  With the McGill Melzack Pain Questionnaire, the location of the pain, the emotion it creates in the individual, its relationship with time, its severity and the level of livable pain for the individual will be determined.
electrogoniometer change | change from baseline electrogoniometer change at 2 weeks
  The range of motion of the cervical region of the individuals participating in the study will be evaluated with an electrogoniometer. This device consists of six axes rotating potentiometers and seven connections. The end joints, which are considered fixed by the strapping system, are fixed at the level of the first thoracic vertebra. The other link is placed on the head with an adjustable helmet. This whole system is very light. It enables the monitoring of three-dimensional continuous and unrestricted neck movements relative to the thorax. The system measures flexion, extension, lateral flexion and rotation.
MyotonPRO device change | change from baseline MyotonPRO device change at 2 weeks
  The muscle tone of the individuals participating in the study will be evaluated with MyotonPRO. MyotonPRO is a portable device that measures muscle tone. It measures the mechanical impulses of the soft tissue with mechanical oscillations. A brief mechanical stimulus is applied to the skin over the muscle, followed by rapid relaxation. It measures the reflective resistance of the muscle to deformation of the applied force in Newtons/meter (N/m). The stiffness value is calculated as the ossification or maximum displacement of the tissue and the maximum acceleration. Larger values indicate a harder muscle. The muscle tone of the upper trapezius, sternocleidomastoid, and suboccipital muscles will be measured.
Flexion endurance test change | change from baseline Flexion endurance test change at 2 weeks
  The endurance of the cervical flexor muscles of the individuals participating in the study will be measured with the craniocervical flexion test using a stabilizer device. People lie on their back in a hooked position. Individuals will then be asked to bring their necks into the chin tuck position and feel the neck position. Subjects will be set to 20 mmHg in the stabilizer device and will be asked to increase these pressures by 2 mmHg until they reach 30 mmHg, stay at each pressure for 30 seconds, and complete the test by giving a 30-second rest period after each pressure. The test will be stopped when the individual is unable to complete the test, is in position, and feels excruciating pain.
Extension endurance test change | change from baseline extension endurance test change at 2 weeks
  In the endurance evaluation of neck extensors, subjects will lie face down on the examination bed with their hands at their sides and their heads will be suspended from the bed until they are at chest level. The two-pound weight will hang just above ear level. With this weight, they will be asked to lift their heads back and not change this position until they get tired. The time they can hold the position will be recorded in seconds.

SECONDARY OUTCOMES:
Headache Impact Scale (HIT-6) change | change from baseline Headache Impact Scale (HIT-6) at 2 weeks
  Headache Impact Scale (HIT-6) will be applied to the individuals participating in the research. This scale consists of 6 items. This scale is used to evaluate how much a headache at work affects school, home and social life. It includes pain, social life, role task, energy, cognitive status, and psychological problems. The Turkish validity and reliability study of the scale was conducted. A score between 36 and 78 can be obtained from this scale. Grade 1: No effect if scale score ≤49, Grade 2: 50-55 moderately affected, Grade 3: 56-59 significantly affected, and Grade 4: ≥60 severely affected.
Corbin Posture Index change | change from baseline Corbin Posture Index at 2 weeks
  Posture analysis will be performed to determine the changes in the posture of the individuals included in the study. These changes will be scored using a form prepared by Corbin et al. that includes lateral and posterior observations. This form does not detect postural disorders by observation made from the two planes mentioned, but is based on scoring according to their severity. Head anterior tilt, rounded back, shoulder protraction, kyphosis, lordosis, abdominal prolapse, genu recurvatum, head lateral tilt, scapula protrusion, and scoliosis will be evaluated. Points will be summed last and postural status will be classified according to the total score. 0-2 points as excellent, 3-4 points as very good, 5-7 points as good, 8-11 points as moderate, >12 points as bad.
The Pittsburgh Sleep Quality Index (PSQI) change | change from baseline The Pittsburgh Sleep Quality Index (PSQI) at 2 weeks
  The Pittsburgh Sleep Quality Index will be made to the participants in the study. PSQI is a scale that provides information about sleep quality and the type and severity of sleep disturbance in the last month. In this scale, the sleep quality of the person; sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleeping pill use, and daytime dysfunction. The Turkish validity and reliability study of the scale was conducted. Each of the questionnaire questions is scored between 0-3, with high scores reflecting poor sleep quality. If the total score obtained from the scale is below 5, it is defined as 'Good sleep quality', and if it is 5 and above, it is defined as 'Poor sleep quality'.

CONTACTS AND LOCATIONS:
Overall Officials: Berrak Varhan, Study Director — İstinyeU
Locations (1):
- Bursa VM Medical Park Hospital, Bursa, Osmangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No